CLINICAL TRIAL: NCT06475417
Title: Phase II Study of Neoadjuvant Adebrelimab, Docetaxel, Oxaliplatin, and S-1 in Patients With Resectable Advanced Gastric Cancer
Brief Title: Neoadjuvant Adebrelimab + DOS in Locally Advanced Resectable Gastric Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tang-Du Hospital (Other)
Collaborators: Jiangsu Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202404-05
Record Dates: First submitted 2024-05-28; First posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Gastric Cancer
Keywords: Gastric Cancer; Resectable; Neoadjuvant; ICIs
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adebrelimab combined with DOS (Experimental): After signing the informed consent, they are screened to meet the inclusion criteria. After receiving the standard dose of adebrelimab combined with DOS regimen for 3 courses of treatment before surgery, and within 3-6 weeks after the completion of the third administration, preoperative imaging examination is used to evaluate the efficacy of new adjuvant treatment and the possibility of radical D2 resection, The patient underwent radical surgical treatment for gastric cancer and observed pCR.
  Interventions: Drug: Adebrelimab combined with DOS

INTERVENTIONS:
Drug: Adebrelimab combined with DOS — After signing the informed consent, they are screened to meet the inclusion criteria. After receiving the standard dose of adebrelimab combined with DOS regimen for 3 courses of treatment before surgery, and within 3-6 weeks after the completion of the third administration, preoperative imaging examination is used to evaluate the efficacy of new adjuvant treatment and the possibility of radical D2 resection, The patient underwent radical surgical treatment for gastric cancer and observed pCR

SUMMARY:
To evaluate the efficacy and safety of adebrelimab combined DOS in neoadjuvant treatment of locally advanced resectable gastric cancer.

DETAILED DESCRIPTION:
This prospective, single-center, single-arm clinical trial aims to enroll 42 treatment-naïve patients diagnosed with locally advanced gastric adenocarcinoma who are deemed operable. Following informed consent, patients will undergo screening to confirm eligibility. Subsequently, eligible participants will receive the standard dosage of Adebrelimab in combination with the DOS regimen for three cycles as neoadjuvant therapy prior to surgery. Within 3-6 weeks after completing the third cycle, preoperative imaging will be conducted to assess the efficacy of the novel neoadjuvant treatment and feasibility of achieving radical D2 resection. Patients will then undergo radical surgical resection for gastric cancer, with pathological complete response (pCR) being observed.

ELIGIBILITY:
Inclusion Criteria:

1. Participants will be recruited voluntarily and will provide informed consent before enrollment. They are expected to demonstrate good compliance and willingness to adhere to the study protocol, including attending follow-up visits as required.
2. Inclusion criteria for participant eligibility are as follows:

1）Age between 18 and 75 years, with no gender restrictions. 2）Histopathological confirmation of locally advanced gastric or gastroesophageal junction adenocarcinoma obtained through gastric endoscopic biopsy.

3）Clinical staging consistent with T2-3N+M0 or T4aNanyM0, confirmed by imaging (CT/MRI) and endoscopic ultrasound.

4）Eastern Cooperative Oncology Group (ECOG) performance status of 0-1. 5）Expected survival of at least 12 weeks. 3.Prior to treatment initiation, participants must meet the following criteria related to vital organ function within the preceding 7 days:

1. Hematological parameters: Hemoglobin (Hb) ≥ 90 g/L, Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L, Platelets (PLT) ≥ 80 × 10^9/L (no recent blood transfusions within 14 days).
2. Biochemical parameters: Total bilirubin (TBIL) ≤ 1.5 × upper limit of normal (ULN), Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) ≤ 2.5 × ULN, Serum creatinine (Cr) ≤ 1.5 × ULN or Creatinine clearance rate (CCr) ≥ 60 ml/min.
3. Doppler ultrasound assessment: Left ventricular ejection fraction (LVEF) ≥ lower limit of normal (50%).

4.Female participants of childbearing potential must agree to use effective contraception during the study and for 6 months after the end of the study period. They must provide negative serum or urine pregnancy tests within 7 days before enrollment and must not be lactating. Male participants must also agree to use effective contraception during the study and for 6 months following its conclusion.

5.All participants must provide voluntary informed consent before participation in the study.

Exclusion Criteria:

1. History of malignancies within the past 5 years, excluding cured cervical carcinoma in situ, non-melanoma skin cancer, and superficial bladder tumors.
2. Patients with tumors invading adjacent organs (e.g., aorta or trachea), posing a high risk of bleeding or fistula formation.
3. Subjects requiring systemic treatment with corticosteroids (>10 mg prednisone or equivalent daily) or other immunosuppressive agents within 14 days prior to study treatment initiation, except for those with no active autoimmune disease who may receive inhaled or topical corticosteroids at doses equivalent to >10 mg prednisone daily or adrenal replacement steroid doses.
4. Patients with significant malnutrition requiring intravenous nutrition or continuous infusion therapy requiring hospitalization. Patients with well-controlled nutrition for ≥28 days before randomization may be included.
5. Participants receiving live vaccines/attenuated vaccines within 30 days after the first treatment.
6. Unresolved toxicities of grade ≥4 as per CTCAE 4.02 due to previous treatments, excluding alopecia and ≤grade 2 neuropathy caused by oxaliplatin.
7. Allergic reactions or contraindications to any study drug components.
8. Patients with severe and/or uncontrolled diseases, including hypertension, myocardial ischemia or infarction, arrhythmias, congestive heart failure, severe or uncontrolled diseases or active infections, renal failure, immunodeficiency diseases, poorly controlled blood glucose, seizures, history of interstitial lung disease, pulmonary fibrosis, or any condition interfering with the detection and management of suspected drug-related toxicities.
9. Patients with current gastrointestinal diseases such as intestinal obstruction or those at risk of gastrointestinal bleeding, perforation, or obstruction.
10. Patients who have undergone surgical treatment, incisional biopsy, or significant traumatic injury within 28 days prior to enrollment.
11. Patients with any bleeding events of grade ≥3 per CTCAE within 4 weeks before enrollment, or those with unhealed wounds, ulcers, or fractures.
12. Participants with thrombotic events (arterial or venous) within 3 months, such as cerebrovascular accidents, deep vein thrombosis, or pulmonary embolism.
13. Subjects planning to undergo or who have previously undergone allogeneic organ or bone marrow transplantation, including liver transplantation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-05-24 (Actual); Primary Completion 2025-05-20 (Estimated); Study Completion 2026-04-26 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate（pCR） | 7 days after surgery
  Pathological complete response rate according to Becker standard

SECONDARY OUTCOMES:
Major pathologic response (MPR) | 7 days after surgery
  MPR is defined as less than 10% residual viable tumor after neoadjuvant therapy.
Disease-free survival（DFS） | Long term follow-up will continue until the death of the subject or the end of the study, at least three years
  The length of time after primary treatment for a cancer ends that the patient survives without any signs or symptoms of that cancer
R0 resection rate | postoperative 6 hours
  Proportion of R0 level surgery performed.
Overall Survival（OS） | Long term follow-up will continue until the death of the subject or the end of the study, at least three years
  Overall survival (OS) refers to the time that researchers evaluate from recording the first chemotherapy to death (of any cause).
Objective response rate（ORR） | 7 days before surgery
  Per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) using Investigator assessments, is defined as the number (%) of patients with response of Complete Response or Partial Response.
Event-free survival（EFS） | Preoperative progression, postoperative recurrence, and death from any cause
  The length of time after primary treatment for a cancer ends that the patient remains free of certain complications or events that the treatment was intended to prevent or delay.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Long term follow-up will continue until the death of the subject or the end of the study, at least three years
  Adverse reactions to chemotherapy and immunotherapy were graded according to the NCI-CTCAE4.0 grading criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Tangdu Hospital Affiliated to the Fourth Military Medical University, Xi'an, Shannxi, China

IPD SHARING:
Plan to Share IPD: No